CLINICAL TRIAL: NCT04625699
Title: A Feasibility Study of Durvalumab + Tremelimumab in Resected Non Small Cell Lung Cancer (NSCLC) Patients With Detectable Circulating Tumor DNA After Adjuvant Treatment
Brief Title: Study of Durvalumab + Tremelimumab in NSCLC Patients After Adjuvant Treatment
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Contract was never finalized.
Sponsor: Catherine Shu (Other)
Responsible Party: Sponsor-Investigator, Catherine Shu, Assistant Professor of Medicine, Columbia University
Organization: Columbia University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAT0800
Record Dates: First submitted 2020-11-06; First posted 2020-11-12 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-06

CONDITIONS: Nonsmall Cell Lung Cancer
Keywords: II-IIIB
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — durvalumab; tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- durvalumab+ tremelimumab (Experimental): durvalumab will be administered Q4weeks and tremelimumab will be administered Q8 weeks
  Interventions: Drug: Durvalumab; Drug: Tremelimumab

INTERVENTIONS:
Drug: Durvalumab — 4 doses of Durvalumab 1500 mg IV Day 1, q28 days (For example, interventions involving drugs may include dosage form, dosage, frequency, and duration.)
  Other Names: MEDI4736, IMFINZI
Drug: Tremelimumab — 2 doses of Tremelimumab 300 mg IV Day 1, q56 days
  Other Names: formerly CP-675,206

SUMMARY:
The purpose of this study is to determine whether it is feasible and safe to give research participants investigational treatment with durvalumab and tremelimumab after they have completed standard treatment for NSCLC and once they have detectable circulating tumor DNA (ctDNA) in the blood before there is evidence of disease recurrence on imaging studies. These investigational agents are a type of immunotherapy, which is a treatment that activates your own body's immune system to treat cancer.

DETAILED DESCRIPTION:
This is an open label, single arm, pilot study of adjuvant durvalumab+ tremelimumab (D+T) for patients with stage II-IIIB (excluding N3) NSCLC.The trial will evaluate the feasibility of adjuvant D+T in patients who have undergone surgical resection and standard of care (SOC) adjuvant treatment and subsequently develop detectable plasma ctDNA. 15 evaluable patients will be enrolled. Patients with resected stage II-IIIB (excluding N3) NSCLC who have completed adjuvant standard of care treatment will be pre-screened and consented for the trial. They will undergo ctDNA testing with the Signatera assay at the completion of adjuvant treatment and every 4 months thereafter with standard CT imaging assessment up to 1 year. Patients with detectable ctDNA at a mutant allele frequency of >0.1% and no evidence of recurrence on CT imaging will be enrolled in the trial. They will receive durvalumab every 4 weeks for 4 cycles and tremelimuamb on cycles 1 and 3 with concomitant plasma ctDNA quantification. Patients will be followed with standard CT imaging of the chest as well as routine and exploratory blood tests every 4 months until 1 year after completion of D+T. They will also be followed for up to 3 years for determination of DFS and OS.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years
* Patients must have pathologically confirmed NSCLC; no mixed NSCLC/SCLC histology allowed
* Stage II-IIIB (8th edition) disease who have undergone surgical resection, excluding patients with N3 disease
* Must have documentation that the tumor does not harbor an activating EGFR mutation, ALK gene rearrangement, or a ROS1 gene rearragement
* Must have adequately recovered from the toxicity and/or complications of surgery prior to initiation of durvalumab+tremelimumab
* Detectable ctDNA at a mutant allele frequency of >0.1% after surgical resection and completion of adjuvant treatment
* No evidence of clinical disease on CT chest/abdomen/pelvis at the time of ctDNA detection
* Completed standard of care adjuvant treatment at least two weeks prior to day 1 of durvalumab+tremelimumab
* Archived tumor tissue: formalin-fixed paraffin-embedded (FFPE) tumor specimens in paraffin block or at least 10 unstained slides, with an associated pathology report.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol. Written informed consent and any locally required authorization (e.g. Health Insurance Portability and Accountability Act) must be obtained from the patient/legal representative prior to performing any protocol-related procedures, including screening evaluations
* Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following agespecific requirements apply:

  * Women <50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and folliclestimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
  * Women ≥50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy). Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Body weight > 30 kg
* Must have a life expectancy of at least 12 weeks
* Ability to comply with the study protocol, in the investigator's judgment
* Adequate organ and marrow function

Exclusion Criteria:

* Concurrent enrollment in another clinical study, unless it is an observational (noninterventional) clinical study or during the follow-up period of an interventional study
* Any concurrent chemotherapy, immunotherapy, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) or herbal therapy is acceptable.
* History of another primary malignancy except for: Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of immune therapy and of low potential risk for recurrence; adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease; adequately treated carcinoma in situ without evidence of disease; malignancy undergoing active surveillance per stand of care management (e.g., chronic lymphocytic leukemia Rai Stage 0, prostate cancer with Gleason score 6, and prostate-specific antigen [PSA] 10 mg/mL, etc.)
* Any unresolved toxicity NCI CTCAE v.5.0 Grade 2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria. Patients with Grade 2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Physician. Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab or tremelimumab may be included only after consultation with the Study Physician.
* Has untreated central nervous system (CNS) metastases and/or carcinomatous meningitis identified either on the baseline brain imaging (RECIST)) for details on the imaging modality) obtained during the screening period or identified prior to signing the ICF
* History of allergic reactions attributed to compounds of similar chemical or biologic
* Patients with active hepatitis B or C infections or a history of HIV infection. These participants will be ineligible due to potential for worsening of infection with the use of immunotherapy. Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
* History of active primary immunodeficiency
* Known clinically significant liver disease, including active viral, alcoholic, or other hepatitis; cirrhosis; fatty liver; and inherited liver disease Known hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion: Patients with vitiligo or alopecia; hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement; any chronic skin condition that does not require systemic therapy; patients without active autoimmune disease in the last 5 years may be included but only after consultation with the study physician; celiac disease controlled by diet alone
* Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, including TB, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent
* Major surgical procedure within 28 days prior to Cycle 1, Day 1 or anticipation of need for a major surgical procedure, excluding lung cancer resection, during the course of the study
* Administration of a live, attenuated vaccine within 30 days before Cycle 1, Day 1 or anticipation that such a live, attenuated vaccine will be required during the study.
* Patients, if enrolled, should not receive live vaccine whilst receiving treatment and up to 30 days after durvalumab, tremelimumab administration.
* History of interstitial lung disease or pneumonitis of any cause
* Pregnant women are excluded from this study because durvalumab and tremelimumab are investigational agents with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with durvalumab and tremelimumab, breastfeeding should be discontinued if the mother is treated with durvalumab and tremelimumab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-12 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Number of evaluable patients enrolled | 36 months
  To assess the feasibility of identifying and recruiting patients for adjuvant treatment with durvalumab+tremelimumab (D+T) in the setting of molecular residual disease based on ctDNA positivity after surgical resection and standard of care treatment for stage II-IIIB NSCLC. The target is a total of 15 with a projected accrual rate of 2-3 patients per month.

SECONDARY OUTCOMES:
ctDNA clearance | 36 months
  To assess the dynamics of ctDNA in response to treatment with adjuvant durvalumab+tremelimumab. This will be reported with 95% confidence intervals based on the exact binomial distribution.
Overall survival | Up to 36 months
  To determine the duration of overall survival with adjuvant durvalumab+tremelimumab
Disease free survival | Up to 36 months
  To determine the duration of disease free survival with adjuvant durvalumab+tremelimumab
Adverse events rate | 36 months
  To evaluate the safety of adjuvant D+T, adverse events will be scored according to NCI CTCAE v5.0 and their frequency and nature will be tabulated by categories. This will be reported with 95% confidence intervals based on the exact binomial distribution.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Shu, MD, Principal Investigator — Columbia University

IPD SHARING:
Plan to Share IPD: No